CLINICAL TRIAL: NCT03811145
Title: A Double-Blind Randomised Placebo-controlled Phase IIb Clinical Trial to Study the Efficacy & Safety of a Novel Platelet Lysate Gel in the Treatment of Lateral Epicondylitis
Brief Title: An Investigation of Tendoncel, a Novel Topical Platelet Lysate Gel, in the Treatment of Lateral Epicondylitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cell Therapy Ltd. (Industry)
Collaborators: George Papanicolaou Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CTL/LE/01/0514
Record Dates: First submitted 2019-01-16; First posted 2019-01-22 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Lateral Epicondylitis
Keywords: Topical; Gel; Platelet; Growth factor; Regenerative
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tendoncel (Experimental): Topically applied experimental gel - Tendoncel. 80ul applied once a day for 21 consecutive days.
  Interventions: Biological: Tendoncel
- Placebo control gel (Placebo Comparator): Placebo control gel. Similar to Tendoncel but without platelet derived small molecules and growth factors. 80ul applied once a day for 21 consecutive days.
  Interventions: Other: Placebo control gel

INTERVENTIONS:
Biological: Tendoncel — Platelet lysate gel
  Arms: Tendoncel
Other: Placebo control gel — Placebo control gel
  Arms: Placebo control gel

SUMMARY:
Current treatments for lateral epicondylitis include: rest, behaviour modification and physiotherapy, anti-inflammatory medication - both steroidal and non-steroidal, and surgery. Current experimental therapies include muscle relaxants to reduce muscle tone and force on the epicondyle, laser therapy to stimulate collagen production, and blood based therapies including the injection of autologous blood and protein rich plasma.

Cell Therapy Ltd (trading as Celixir) has developed a regenerative gel that combines isolated allogeneic platelet growth factors and a cellulose-derivative gel.

DETAILED DESCRIPTION:
Lateral epicondylitis, also called "tennis elbow" is a common condition affecting 1 to 3% of the population; most commonly individuals aged 35 to 55 years. It is frequently self limiting but can lead to refractory symptoms in a minority of cases. Pain is localised to the lateral epicondyle of the elbow at the point of insertion of the common extensor tendon. Although associated with repetitive movement of the extensor muscles of the forearm, frequently no precipitating cause can be discerned.

The term "epicondylitis" is a misnomer as histological investigations have revealed that there is only limited inflammation, and the term "epicondylosis" should be employed, due to the degenerative nature of the condition.

The condition is divided in to 4 stages, though progression may not occur through all four. Firstly, there is acute inflammation that is quick to resolve. Secondly, prolonged injury results in an increase in fibroblasts, vascular hyperplasia, disorganised collagen disposition and degeneration of the tendon. Thirdly, further accumulation of structural alterations leads to partial or complete tendon rupture. Stage 4 exhibits the same features as 2 and 3 but with the addition of calcification.

Current treatments for lateral epicondylitis include: rest, behaviour modification and physiotherapy, anti-inflammatory medication both steroidal and non-steroidal, and surgery. Current experimental therapies include muscle relaxants to reduce muscle tone and force on the epicondyle, laser therapy to stimulate collagen production, and blood based therapies including the injection of autologous blood and protein rich plasma. Trials of the latter two treatments give conflicting results due to variations in protocol and trial design.

Cell Therapy Ltd has developed a regenerative gel, Tendoncel, that combines isolated platelet growth factors and cellulose-derivative gel. Tendoncel consists of a proprietary platelet lysate formulation that is easy to apply to the skin.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years and over and in good general health
* Subjects who have a diagnosis of lateral epicondylitis, Cozen's test
* Subjects who are willing to attend all study assessments and follow-up appointments
* Subjects who are able to understand the study, and are willing to co-operate with the study procedures and restrictions

Exclusion Criteria:

* Subjects have been receiving additional concurrent treatment (e.g. surgical or steroid injection) for lateral epicondylitis.
* Subjects who have medial epicondylitis or another condition of the elbow (test side only)
* Subjects who have participated in any clinical study during the previous 30 days of initiation of this study
* Subjects with a history of alcohol, substance or drug abuse in the previous 12 months
* Subjects with any significant concurrent illness
* Subjects with a heart pacemaker
* Subjects with diabetes either type I or type II (owing to possible poor wound healing)
* Subjects that have undergone surgery in the past 3 months
* Subjects with any active or significant history of skin disorders at the treatment area(s) e.g. hypo pigmentation (vitiligo)
* Subjects with any inflammatory skin condition (eczema, psoriasis, herpes simplex/complex)
* Subjects with a history (or family history) of skin cancer, skin tumours or any other malignant disease
* Subjects with any irritation, tattoo's, piercings, scars, birthmarks, or heavy presence of freckles at the treatment site(s)
* Subjects currently taking anti-histamine or steroid medication
* Subject who due to impaired mobility would not be able to undertake independent care
* Subjects who are pregnant or who are breast feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire | Baseline
  15 question questionnaire measuring pain and function. Total scores from 15 questions compared - pain and function combined. Scale: 10 to 100 (best to worst). Difference between test and control scores compared.
Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire | Day 23 (end of treatment).
  15 question questionnaire measuring pain and function. Total scores from 15 questions compared - pain and function combined. Scale: 10 to 100 (best to worst). Difference between test and control scores compared.
Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire | 4 weeks follow up
  15 question questionnaire measuring pain and function. Total scores from 15 questions compared - pain and function combined. Scale: 10 to 100 (best to worst). Difference between test and control scores compared.
Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire | 6 weeks follow up.
  15 question questionnaire measuring pain and function. Total scores from 15 questions compared - pain and function combined. Scale: 10 to 100 (best to worst). Difference between test and control scores compared.
Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire | 3 months follow up.
  15 question questionnaire measuring pain and function. Total scores from 15 questions compared - pain and function combined. Scale: 10 to 100 (best to worst). Difference between test and control scores compared.
Patient-Rated Tennis Elbow Evaluation (PRTEE) questionnaire | Mean of 47 weeks follow up.
  15 question questionnaire measuring pain and function. Total scores from 15 questions compared - pain and function combined. Scale: 10 to 100 (best to worst). Difference between test and control scores compared.
Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Baseline
  30 question questionnaire measuring disabilities of the upper limb. Scale from 0 to 100 (best to worst). Difference between test and control scores compared.
Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Day 23.
  30 question questionnaire measuring disabilities of the upper limb. Scale from 0 to 100 (best to worst). Difference between test and control scores compared.
Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | 4 week follow up.
  30 question questionnaire measuring disabilities of the upper limb. Scale from 0 to 100 (best to worst). Difference between test and control scores compared.
Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | 6 week follow up.
  30 question questionnaire measuring disabilities of the upper limb. Scale from 0 to 100 (best to worst). Difference between test and control scores compared.
Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | 3 months follow up
  30 question questionnaire measuring disabilities of the upper limb. Scale from 0 to 100 (best to worst). Difference between test and control scores compared.
Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Mean of 47 weeks follow up.
  30 question questionnaire measuring disabilities of the upper limb. Scale from 0 to 100 (best to worst). Difference between test and control scores compared.
Pain free grip strength | Baseline
  Measured using a dynamometer. Results compared between test and control elbows, and between study and contralateral elbow (internal control).
Pain free grip strength | Day 23
  Measured using a dynamometer. Results compared between test and control elbows, and between study and contralateral elbow (internal control).
Pain free grip strength | Mean of 47 weeks follow up (final follow up).
  Measured using a dynamometer. Results compared between test and control elbows, and between study and contralateral elbow (internal control).

SECONDARY OUTCOMES:
Safety - Number of participants in each group with adverse events. | Day 3 (1st treatment visit), day 7, day 14, day 21, day 23 (end of treatment). Follow ups: 4 weeks, 6 weeks, 3 months and mean of 47 weeks.
  Measured by participant questionnaire. Comparison of the number of participants in each group with cutaneous events - "redness", "rash", "swelling" or changes at gel site. Classed as none, mild, moderate or severe. Plus any other event mentioned by the participants.
Safety: Immune response - blood IgE levels. Difference between test and control groups. | Baseline
  Measurement of blood IgE levels. Test and control averages compared. Normal is <100IU/mL.
Safety: Immune response - blood IgE levels. Difference between test and control groups. | Day 7
  Measurement of blood IgE levels. Test and control averages compared. Normal is <100IU/mL.
Safety: Immune response - blood IgE levels. Difference between test and control groups. | Day 23
  Measurement of blood IgE levels. Test and control averages compared. Normal is <100IU/mL.
Safety: Immune response - blood IgE levels. Number of participants in each group with a normal baseline reading and a subsequently elevated reading. | Baseline, day 7 and day 23.
  Measurement of blood IgE levels. Comparison of the number of participants in each group, test and control, with a normal baseline reading of blood IgE and a subsequently elevated IgE reading. Normal is <100IU/mL.

CONTACTS AND LOCATIONS:
Overall Officials: Givissis Panagiotis, MD, Principal Investigator — Aristotle University of Thessaloniki, General Hospital of Papanikolaou
Locations (1):
- Orthopaedic Clinic of Aristotle University of Thessaloniki, General Hospital of Papanikolaou, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad Z, Siddiqui N, Malik SS, Abdus-Samee M, Tytherleigh-Strong G, Rushton N. Lateral epicondylitis: a review of pathology and management. Bone Joint J. 2013 Sep;95-B(9):1158-64. doi: 10.1302/0301-620X.95B9.29285. PMID 23997125
- See also: Ahmad et al., (2013) — https://online.boneandjoint.org.uk/doi/pdf/10.1302/0301-620X.95B9.29285